CLINICAL TRIAL: NCT01013051
Title: Effect of Gastric Bypass on the Absorption of Metformin
Acronym: ABSORB-Met
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Raj Padwal, University of Alberta
Other Study IDs: RES0002122
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-03

CONDITIONS: Obesity; Gastric Bypass
Keywords: obesity; gastric bypass; metformin; pharmacokinetics; absorption
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Post Gastric Bypass
- Obese Controls: age, BMI, gender matched

SUMMARY:
Background: Gastric bypass is the most commonly performed type of bariatric (obesity) surgery, has dramatically increased in popularity and is now considered to be preferred treatments in severely obese patients that fail non-surgical therapy - particularly in patients with type 2 diabetes. Drug malabsorption is a potential concern post-gastric bypass because intestinal length is reduced.

Purpose: The purpose of this controlled, pharmacokinetic study is to determine whether the absorption of a single dose of metformin, the first line drug treatment in patients with type 2 diabetes, is significantly reduced after gastric bypass.

Methods: A single dose of standard release metformin 1000 mg will be administered to patients who have undergone gastric bypass and to patients who have not received surgery but are on the wait list (wait-listed controls). Blood sampling and urine sampling will occur in standardized fashion over the ensuing 24 hours to measure and compare the absorption of metformin between study arms. 34 patients total will be recruited.

Significance: Following completion of this study, we will better understand how gastric bypass affects metformin absorption. Ultimately, this information will help to ensure that this patient population is receiving optimal doses of this important drug treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients living within and around Edmonton that have been referred to the Alberta Health Services Weight Wise Program

Exclusion Criteria:

1. Undergone or undergoing revision of a previous bariatric procedure
2. Any major post-operative gastrointestinal complications, such as an anastomotic leak, outlet obstruction or persistent vomiting
3. Currently on metformin therapy
4. Any contraindications to metformin therapy such as:

   1. allergy to the drug
   2. chronic metabolic acidosis
   3. history of lactic acidosis
   4. liver failure or baseline liver enzymes higher than 3-fold above the upper limit of normal
   5. congestive heart failure
   6. renal failure (glomerular filtration rate < 60 ml/min)
   7. alcoholism
   8. acute illness
   9. fatty liver disease
5. Pregnant or nursing
6. Not taking furosemide or nifedipine (both drugs may increase metformin absorption by 15-20%)the day of visit 2.
7. Any other medical, social or geographic condition, which, in the opinion of the investigator would not allow safe completion of the study protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Post gastric bypass and obese controls
  1. Male and Female
  2. 18 - 60 years old
  3. ≥ 3 months post-RYGB surgery or wait listed for bariatric surgery
  4. Able to provide written informed consent.
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2009-09; Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Area-under-the-curve of metformin absorption (0-infinity) | cross-sectional

SECONDARY OUTCOMES:
AUC (0-24h) | cross-sectional
tmax | cross-sectional
cmax | cross-sectional
AUC glucose (0-8h) | cross-sectional
bioavailability of metformin (urine metformin concentration from 0-infinity) | cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Raj Padwal, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital Clinical Investigation Unity, Edmonton, Alberta, Canada